CLINICAL TRIAL: NCT02840526
Title: Thoracic Paravertebral Block in Postoperative Pain Management After Renal Surgery
Brief Title: Thoracic Paravertebral Block in Pain Management After Renal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Silesian University of Medicine (Other)
Responsible Party: Principal Investigator, Maja Copik, M.D., Silesian University of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUM-PSK-1
Record Dates: First submitted 2013-11-22; First posted 2016-07-21 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Postoperative Pain
Keywords: PVB; PCA; nephrectomy; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — cisatracurium; Sevoflurane; Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PVB group (Experimental): Thoracic paravertebral blockade PVB (preoperatively) Bupivacaine WZF Sopodorm Propofol WZF Fentanyl WZF Nimbex Sevorane Intubation Oxynorm Ketonal Paracetamol Kabi
  Interventions: Procedure: Paravertebral blockade (PVB); Drug: Sopodorm; Drug: Propofol WZF; Drug: Nimbex; Drug: Fentanyl WZF; Drug: Sevorane; Device: Intubation; Drug: Oxynorm; Drug: Paracetamol Kabi; Drug: Ketonal; Drug: Bupivacaine WZF
- GEN group (Other): Sopodorm Propofol WZF Fentanyl WZF Nimbex Sevorane Intubation Oxynorm Ketonal Paracetamol Kabi
  Interventions: Drug: Sopodorm; Drug: Propofol WZF; Drug: Nimbex; Drug: Fentanyl WZF; Drug: Sevorane; Device: Intubation; Drug: Oxynorm; Drug: Paracetamol Kabi; Drug: Ketonal

INTERVENTIONS:
Procedure: Paravertebral blockade (PVB) — preoperative ThPVB performed unilaterally at Th10 level
  Arms: PVB group
Drug: Sopodorm — midazolam 0,1 mgkg-1 intravenously (anesthesia induction)
Drug: Propofol WZF — propofol 2 mgkg-1intravenously (anesthesia induction)
Drug: Nimbex — cis-atracurium 0,15 mgkg-1 intravenously (anesthesia induction)
Drug: Fentanyl WZF — fentanyl 1,5 µgkg-1 intravenously (anesthesia induction)
Drug: Sevorane — sevoflurane in 1 MAC (Minimal Alveolar Concentration) - anesthesia maintenance
Device: Intubation — Intratracheal intubation with a single lumen endotracheal tube
Drug: Oxynorm — 1 mgml-1 concentration oxycodone solution intravenously
Drug: Paracetamol Kabi — 1g paracetamol intravenously every 6 hours
Drug: Ketonal — 100 mg ketoprofen intravenously every 12 hours
Drug: Bupivacaine WZF — 0,3 ml kg-1 0,5% plain bupivacaine (regional anesthesia - paravertebral blockade)
  Arms: PVB group

SUMMARY:
Objective: The objective of the study was to assess the usefulness of ThPVB in postoperative pain management after open renal resection surgery.

Design, setting, participants: It was a prospective, randomised, open label study held in a university hospital between 08.2013-12.2014. 58 Patients enrolled in the study were scheduled for elective open renal surgery (open nephrectomy or open nephron-sparing surgery) and randomised into two groups - group PVB (n=27) and group GEN (n=31).

Interventions: PVB group received preoperative ThPVB with 0,5% bupivacaine followed by general anaesthesia. GEN group received standard general anaesthesia. Both groups were treated postoperatively with oxycodone IV PCA (patient controlled analgesia) combined with non-opioid analgesics as rescue drugs. The investigators recorded pain severity in VAS, oxycodone requirement in time points, total oxycodone requirement, and sedation levels throughout the first 48h. The investigators measured opioid related adverse events 24 and 48 h postoperatively and patients satisfaction 48h postoperatively.

DETAILED DESCRIPTION:
In PVB group before the induction of general anaesthesia a single shot thoracic paravertebral blockade was performed. ThPVB was performed on Th7-Th10 level, approximately 2,5 - 3 cm lateral from the top of the spinous process with prior ultrasound control of the depth of the transverse process and the pleura. To make the procedure safer the investigators used peripheral nerve stimulation with an isolated 10 cm needle with a start current of 2,5 mA. The needle was inserted until visible muscle activity from intercostal muscles appeared, with a current of 0,5-0,3mA (paravertebral space identification). Next 0,3 ml kg-1 0,5% plain bupivacaine was injected after negative aspiration for air and blood. The efficacy of the blockade was checked after 20 minutes with cold saline.

In both groups, PVB and GEN general anaesthesia was induced with midazolam 0,1 mgkg-1, propofol 2 mgkg-1, cis-atracurium 0,15 mgkg-1 and fentanyl 1,5 µgkg-1. Patients were intubated with a standard single lumen tracheal tube. Anaesthesia was maintained with 1 MAC (Minimal Alveolar Concentration) sevoflurane. For surgical analgesia the investigators used fractional doses of fentanyl 1-3 mg kg-1 if HR (heart rate) or MBP (mean blood pressure) raised above 20% of basal values. Waking up from anaesthesia was in a post-anaesthesia care unit.

Postoperative pain management schedule was identical in both groups. After the surgery, if pain appeared, the patient was given oxycodone i.v. titrated to achieve acceptable analgesia level or until side effects appeared. Every patient received a PCA (Patient controlled analgesia) device with a 1 mgml-1 concentration oxycodone solution with a programmed single bolus dose of 1 mg and a lockout time of 5 minutes. Additionally, patients were given 1g i.v. paracetamol every 6 hours and 100 mg of i.v. ketoprofen every 12 hours.

For 48 h postoperatively, the investigators monitored HR, SBP (systolic blood pressure) , DBP (diastolic blood pressure), sedation level in Ramsay scale, pain intensity at rest in VAS (visual analogue score) scale, oxycodone requirement in pre-selected time points and total oxycodone requirement. The investigators also recorded opioid-related adverse events 24 and 48 h postoperatively in OBAS scale and patients' satisfaction regarding postoperative analgesia 48 h postoperatively in Likert scale.

ELIGIBILITY:
Inclusion criteria:

* Age 18-75
* Scheduled for elective open nephrectomy or NSS
* Gave written consent
* BMI 19-30
* ASA status I-III

Exclusion criteria:

* Presence of chronic pain
* Chronic mental conditions (depression)
* Contraindications for PVB
* Chest or spine deformations
* Infection in planned site of PVB
* Allergies for drugs used in the study
* Cancer invading chest wall

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Difference in total amount of oxycodone needed in 48 hours after surgery | 48 hours postoperatively

SECONDARY OUTCOMES:
Difference in prevalence of opioid related adverse events in OBAS scale | 24 hours, 48 hours after surgery
Difference in pain level in VAS scale | 48 hours postoperatively
Difference in level of sedation assessed in Ramsay scale | 48 hours after surgery
Difference in patient satisfaction level assessed in Likert scale | 48 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Misiolek, MD PhD, Study Chair — Medical School of Silesia
Locations (1):
- Samodzielny Publiczny Szpital Kliniczny nr 1 SUM Zabrze, Zabrze, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Copik M, Bialka S, Daszkiewicz A, Misiolek H. Thoracic paravertebral block for postoperative pain management after renal surgery: A randomised controlled trial. Eur J Anaesthesiol. 2017 Sep;34(9):596-601. doi: 10.1097/EJA.0000000000000673. PMID 28731925